CLINICAL TRIAL: NCT03350087
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation and Virtual Cycling Training on Upper Limb Function in Patients With Stroke
Brief Title: Efficacy of rTMS and VCT on Upper Limb Function in Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 104-8816A3
Record Dates: First submitted 2017-09-07; First posted 2017-11-22 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Vascular Accident
Keywords: repetitive transcranial magnetic stimulation; stroke; optimal treatment protocol; VR-based cycling training (VCT); randomized controlled trial; motor control; clinical predictors
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- iTBS group (Experimental): In intermittent theta burst stimulation (iTBS group), they received iTBS (80% of active motor threshold) on affected hemisphere.
  Interventions: Device: intermittent theta burst stimulation
- cTBS group (Experimental): In continuous theta burst stimulation (cTBS group), they received cTBS (80% of active motor threshold) on unaffected hemisphere.
  Interventions: Device: continuous theta burst stimulation
- iTBS+cTBS group (Experimental): Continuous theta burst stimulation (cTBS group) at first followed by intermittent theta burst stimulation (iTBS group).
  Interventions: Device: iTBS+cTBS group
- sham TBS group (Sham Comparator): In sham theta burst stimulation (sham TBS group), they received sham TBS stimulation.
  Interventions: Device: sham theta burst stimulation
- VCT group (Experimental): VCT group received the VCT training in addition to traditional rehabilitation. Each UE VCT session involved upper limb cycling training followed by UE training in addition to home program. The cycling program consisted of a warm-up exercise, twenty repetitions of hand push-up movements in the sitting position, UE cycling, and a cool-down exercise.
  Interventions: Device: VCT
- VCT+optimal rTMS group (Experimental): VCT+optimal rTMS group received the VCT training and optimal rTMS in addition to traditional rehabilitation.
  Interventions: Device: VCT+optimal rTMS group

INTERVENTIONS:
Device: intermittent theta burst stimulation — In intermittent theta burst stimulation pattern (iTBS) will intermittently give a 2 s train of TBS every 10s repeated 2 times for a total of 40 times (low pulse: 1200 pulses in total)
  Other Names:
  intermittent theta burst stimulation
  Arms: iTBS group
Device: continuous theta burst stimulation — In continuous burst stimulation pattern (cTBS) will intermittently give a cTBS treatment consists of a continuous train of TBS for 40 seconds repeated for 2 times(low pulse: 1200 pulses in total).
  Other Names:
  continuous burst stimulation
  Arms: cTBS group
Device: iTBS+cTBS group — In iTBS+cTBS pattern, continuous cTBS will be followed by intermittent iTBS (low pulse; 1200 pulses in total)
  Arms: iTBS+cTBS group
Device: sham theta burst stimulation — In sham burst stimulation pattern (sham TBS) will intermittently give a sham TBS treatment consists of a continuous train of TBS for 40 seconds(almost no pulse: 1200 pulses in total).
  Other Names:
  sham theta burst stimulation
  Arms: sham TBS group
Device: VCT — The UE VCT programs were conducted three times per week, for 12 weeks. Each UE VCT session involved upper limb cycling training followed by UE training in addition to home program. The cycling program consisted of a warm-up exercise, twenty repetitions of hand push-up movements in the sitting position, UE cycling, and a cool-down exercise. The warm-up and cool-down exercises involved stretching and relaxing the head, neck, and the upper and lower body.
  Other Names:
  The upper extremity programs virtual cycling training program
  Arms: VCT group
Device: VCT+optimal rTMS group — In VCT+optimal rTMS group, VCT will be combined with optimal rTMS, which has the best outcome in phase 1.
  Arms: VCT+optimal rTMS group

SUMMARY:
Stroke is the major cause of motor impairment and physical disabilities in the adult population. Spasticity and loss of dexterity are the common problems in stroke. Recently, current interventions, such as cycling training, virtual reality (VR) and repetitive transcranial magnetic stimulation (rTMS), were used for the treatment of upper extremity (UE) dysfunction in patients with stroke. However, few studies investigated the effects of the combinations of different treatment strategies using by integrating brain imaging and motor control studies. This project proposes different novel treatment strategies in the treatment of UE dysfunction in patients with stroke: combined inhibitory/facilitatory rTMS, VR-based cycling training (VCT), and combined rTMS and VCT. We hypothesize that the treatment effect of the combined protocol (optimal rTMS protocol and VCT) is more effective than single treatment due to integration of central and peripheral effects. Different treatment protocols will induce different changes in the brain reorganization and motor control, which further improve motor function, activity, participation, and health related quality of life (HRQOL).

DETAILED DESCRIPTION:
This study aims to 1. identify the immediate effects of different treatment protocols in for UE training in these patients through brain image, motor control and clinical measures; 2. to determine the maintaining therapeutic effects; 3. to elucidate the most optimal treatment protocols; 4. to determine the neuro-motor control mechanism underlying clinical improvement; 5. to determine the clinimetric properties of the brain imaging and motor control measure that are responsive and valid for detecting changes after treatment protocol intervention, and 6. to identify clinical predictors influencing the outcome for treatment protocols.

The research will offer valuable motor control biomarkers for outcome prediction and targeting patients who benefit from new protocols. This project is significant for the translational and evidence-based medicine on stroke neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* first stroke
* chronic stroke (onset > 3 months)
* unilateral cerebral lesion with hemiparesis or hemiplegia
* age of 20-80 years
* no epileptic spikes on the EEG

Exclusion Criteria:

* brain stem or cerebellum stroke
* epilepsy
* aneurysm
* arteriovenous malformation
* psychiatric disease
* degenerative disease
* severe cognitive and communicative impairment or aphasia
* severe medical disease
* active medical problems
* metal implant in the body
* pregnancy
* poor cooperation with assessments

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2022-02-11 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of mechanical measurement for stroke after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Kinematic analysis for upper limb
Change from baseline of severity for stroke after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Brunnstrom stage classification(by severity from stage 1 to stage 6), Modified Ashworth Scale (tension of upper limb from min(0) to max (4)) and National Institute of Health Stroke Scale (severity from min(0) to max(4))
Change from baseline of Muscle tone measurement for stroke after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Muscle tone
Change from baseline of Muscle strength measurement for stroke after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Muscle strength

SECONDARY OUTCOMES:
Change from baseline of body composition for stroke in after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  InBodyS10 Body Composition Analyzer
Change from baseline of activity for stroke in after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Barthel Index
Change from baseline of ABAS for stroke in after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Adaptive behavior assessment system
Change from baseline of quality of life for stroke in after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Stroke Impact Scale
Change from baseline of WMFT for stroke in after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Wolf motor function test
Change from baseline of MAL for stroke in after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Motor activity log
Change from baseline of TUG for stroke in after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Timed 'Up & Go' test
Change from baseline of FIM for stroke in after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Functional Independence Measure
Change from baseline of participation for stroke in after 3 weeks treatment and 3 months follow-up | baseline, after 3 weeks of treatment, 3 months
  Nottingham Health Profile

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD, PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen YH, Chen CL, Huang YZ, Chen HC, Chen CY, Wu CY, Lin KC. Augmented efficacy of intermittent theta burst stimulation on the virtual reality-based cycling training for upper limb function in patients with stroke: a double-blinded, randomized controlled trial. J Neuroeng Rehabil. 2021 May 31;18(1):91. doi: 10.1186/s12984-021-00885-5. PMID 34059090